CLINICAL TRIAL: NCT05806671
Title: A Phase II, Single Arm, Open-label Trial of Dalpiciclib Plus Fulvestrant With Pyrotinib in Hormone Receptor-positive, HER2-low Advanced Breast Cancer That Progressed on Previous CDK4/6i Plus AI Therapy
Brief Title: Dalpiciclib Plus Fulvestrant With Pyrotinib in Hormone Receptor-positive, HER2-low Advanced Breast Cancer That Progressed on Previous CDK4/6i Plus AI Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-II-086
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — dalpiciclib; pyrotinib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dalpiciclib, Fulvestrant With Pyrotinib (Experimental): Pyrotinib 320mg/day Dalpiciclib 125 mg/day Fulvestrant 500mg
  Interventions: Drug: Dalpiciclib; Drug: Pyrotinib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Dalpiciclib — Dalpiciclib 125 mg/day orally continuously dosed for 3 weeks followed by 1 week off
  Other Names: SHR6390
Drug: Pyrotinib — Pyrotinib 320mg/day orally continuously
Drug: Fulvestrant — Fulvestrant 500mg intramuscularly on Days 1 and 15 of Cycle 1, and then on Day 1 of each subsequent 28 day cycle

SUMMARY:
The purpose of this study is to determine if the triplet combination of dalpiciclib, fulvestrant, and pyrotinib is safe and effective in the treatment of hormone receptor-positive, HER2-low locally advanced/metastatic breast cancer following treatment with an aromatase inhibitor plus a CDK4/6 inhibitor (palbociclib abemaciclib or ribociclib).

The study will employ a Bayesian Optimal Phase II (BOP2) design which explicitly controls the type I error rate, thereby bridging the gap between Bayesian designs and frequentist designs, and has favorable operating characteristics with higher power and lower risk of incorrectly terminating the trial than some existing Bayesian phase II designs.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women at least 18 years of age with histologically or cytologically confirmed adenocarcinoma of the breast with unresectable or metastatic disease.
2. Most recent tumor biopsy or surgical resection specimen must be either estrogen-receptor (ER) positive, progesterone receptors (PgR) positive, or both, as defined by immunohistochemistry (IHC) ≥1% (as per the American Society of Clinical Oncology (ASCO)-College of American Pathologists (CAP) guidelines).
3. HER2-low breast cancer defined as IHC 2+/ISH- or IHC 1+ (ISH- or untested). (as per the ASCO-CAP guidelines).
4. Postmenopausal status or receiving ovarian ablation with a GnRH agonist such as goserelin. Postmenopausal status is defined by any one of the following criteria:

   * Prior bilateral oophorectomy.
   * Age ≥60 years.
   * Age <60 and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifen, or ovarian suppression) and FSH, LH, and estradiol in the postmenopausal range per local normal If the patient does not meet criteria for postmenopausal status but is receiving ovarian ablation therapy with a gonadotropin-releasing hormone (GnRH) agonist such as goserelin, the patient is eligible for this study, provided that the GnRH agonist is started at least 2 weeks prior to C1D1 of anti-estrogen therapy.
5. Patient must have either measurable disease by RECIST 1.1 or only bone lesions in absence of measurable disease.
6. Eastern Cooperative Group (ECOG) performance status of 0 or 1.
7. Previously treated on CDK 4/6 inhibitor(palbociclib, abemaciclib or ribociclib) with AI for at least 6 months
8. Adequate bone marrow and organ function.

Exclusion Criteria:

1. Patient with symptomatic visceral disease or any disease burden.
2. Patient has received more than one line of chemotherapy for advanced disease.
3. Previous treatment with Dalpiciclib /Pyrotinib /ADCe for advanced disease.
4. Progressed on more than one CDK 4/6 inhibitor
5. Patients with persistent symptoms and unstable brain metastases;
6. Any condition that makes the patient ineligible for endocrine therapy per the investigator's best judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) as Assessed by the Investigator | From start date to date of first documentation of progression or death (assessed up to 12 months)
  Progression free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From start date to date of first documentation of progression or death (assessed up to 12 months)
  Evaluation of disease will be made according to RECIST criteria (version 1.1) in patients with measurable disease. As this study will enroll patients with measureable and un-measurable disease as defined by RECIST v1.1, ORR will only be assessed in evaluable patients. Response rates will be estimated as the proportion of enrolled patients who achieve complete or partial response rate.
Clinical Benefit Rate (CBR) | From start date to date of first documentation of progression or death (assessed up to 12 months)
  Clinical Benefit Rate (CBR) is defined as the percentage of participants with a complete response (CR) or partial response (PR) or with stable disease (SD) as per Response Evaluation Criteria in Solid Tumors (RECIST) V1.1 or Non-Complete Response or Non-Progressive Disease (NCRNPD) during first 24 weeks of first dose. CR=disappearance of all non-nodal target lesions, PR=at least a 30% decrease in the sum of diameter of all target lesions, SD=neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease (PD), PD=at least a 20% increase in the sum of diameter of all target lesions.
Overall Survival (OS) | From start date to date of death (assessed up to 24 months)
  Overall survival is the time from date of first treatment to the date of death due to any cause. If a patient is not known to have died, survival will be censored at the last date of contact.
Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs; All Causalities) | From the signing of the informed consent until 28 days after the last dose of study medication up to 14 months
  An AE is any untoward medical occurrence in a clinical investigation patient administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. An SAE is any untoward medical occurrence at any dose that results in death; is life-threatening; requires hospitalization; results in persistent or significant disability or in congenital anomaly/birth defect. Severity will be graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No